CLINICAL TRIAL: NCT03557424
Title: BEFORE-Study for the Evaluation of Safety and Efficacy of Polyglucosamin and Glucomannan Combination.
Brief Title: BEFORE Study, Efficacy of Refigura
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Heilpflanzenwohl AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BEFORE-Study
Record Dates: First submitted 2018-05-22; First posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Overweight and Obesity; Weight Loss; Efficacy, Self
Keywords: Polyglucosamine; Glucomannan; Weight reduction; Weight loss; without change in lifestyle
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: Three armed, parallel, double blind, Placebo-controlled, interventional study
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blind, randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Polyglucosamine Glucomannan normal dose (Experimental): Patients received the single dose Polyglucosamine und Glucomannan (0,5 g resp. 1 g per Stick) three times per day over 65 days. The drug is administered as a powder which is dissolved in water. The solution is taken orally.
  Interventions: Drug: Polyglucosamine Glucomannan normal dose (Verum)
- Polyglucosamine Glucomannan high dose (Experimental): Patients received the higher dose of Polyglucosamine und Glucomannan (1 g resp. 1,34 g per Stick) three times per day over 65 days. The drug is administered as a powder which is dissolved in water. The solution is taken orally.
  Interventions: Drug: Polyglucosamine Glucomannan high dose (Verum)
- Placebo (Placebo Comparator): Patients received Placebo three times per day over 65 days. The Placebo is administered according to the respective Intervention (Drug: Placebo Comparator: Placebo) as a powder which is dissolved in water. The solution is taken orally.
  Interventions: Drug: Placebo Comparator: Placebo

INTERVENTIONS:
Drug: Polyglucosamine Glucomannan normal dose (Verum) — Patients received Verum three times a day for 65 days. The patients had to dissolve the powder included in one sachet in 250 ml water and drink the solution 15 minutes before each meal. It was recorded whether the patients changed their Lifestyle (their dietary habits and doing sports) during the study.
  Other Names: Polyglucosamine Glucomannan normal dose
  Arms: Polyglucosamine Glucomannan normal dose
Drug: Polyglucosamine Glucomannan high dose (Verum) — Patients received Verum 2 three times a day for 65 days. The patients had to dissolve the powder included in one sachet in 250 ml water and drink the solution 15 minutes before each meal. It was recorded whether the patients changed their Lifestyle (their dietary habits and doing sports) during the study.
  Other Names: Polyglucosamine Glucomannan high dose
  Arms: Polyglucosamine Glucomannan high dose
Drug: Placebo Comparator: Placebo — Patients received Placebo three times a day for 65 days. The patients had to dissolve the powder included in one sachet in 250 ml water and drink the solution 15 minutes before each meal. It was recorded whether the patients changed their Lifestyle (their dietary habits and doing sports) during the study.
  Arms: Placebo

SUMMARY:
The BEFORE study ((B) EFficacy Of REfigura) is designed to demonstrate the efficacy of REFIGURA®. It is a double-blind, randomized, monocentric study.

DETAILED DESCRIPTION:
Core data from the BEFORE study:

Sponsor: Heilpflanzenwohl AG Product: REFIGURA® Title: BEFORE study: Demonstrating the efficacy of REFIGURA® through a double-blind, three-arm, randomized, monocentric study Study duration: 8 weeks (56 days) Study location: MIT Gesundheit GmbH, Stechbahn 20-22, 47533 Kleve CRO: MIT Health GmbH, Stechbahn 20-22, 47533 Kleve Number of study participants: 165 (55 patients per treatment arm)

Summary:

REFIGURA® (manufactured by KITOZYME, Parc Industriel des Hauts-Sarts, Zone 2, Rue de Milmort, 680, BE-4040 Herstal, Belgium, Distribution: Heilpflanzenwohlkraft GmbH), is an approved medical device containing a combination of chitosan (a polyglucosamine ) and glucomannan. Chitosan is a vegetable fiber that binds fats in the intestinal lumen. Both substances are already approved and show few side effects. They are not absorbed into the body, but work directly in the intestine.

The investigational medicinal products are used to treat obesity (weight loss) and to control weight. The effect is based on a reduction in caloric intake, by increasing the feeling of satiety and at the same time the appetite is reduced. As a result, the amount of food consumed is reduced and excessive food (cravings attacks) is prevented. It also reduces the intake of dietary fats.

The study compares three treatment arms:

1. placebo
2. Verum (in the normal, approved dose)
3. Verum (in the double dose)

The patients are weighed, their body fat content is measured and the body size is measured. All measurement methods are non-invasive.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-50 years
* Body mass index (BMI) ≥ 30 kg/m² or
* BMI between 25 and ˂ 30 kg/m² and simultaneous existence of at least one of the following factors:

  1. Overweight-related health disorder (e.g. Hypertension, type 2 Diabetes m.)
  2. Abdominal Obesity
  3. A disease aggravated by obesity
  4. High psychosocial pressure of suffering

Exclusion Criteria:

* Pregnancy (examination with the help of a pregnancy test using urine Lab Test at V2) and lactation
* Alcohol, drugs and drug abuse
* Limited compliance (pre-questionnaire examination)
* History of malignant tumors
* (chronic) Inflammatory diseases of the gastrointestinal tract
* Gastroparesis (stomach paralysis) in the anamnesis
* Signs of an intestinal closure (arising or existing mechanical or paralytic Ileus) in the anamnesis
* Gastric bridging surgery or gastric reduction
* Hypersensitivity or allergy to the ingredients
* Untreated or inadequately treated hypertension
* Diabetes mellitus (examination with the help of a urine tests)
* Treatment with diuretics or insulin
* Cortisone, which has a systemic effect
* Smokers who want to start weaning during the trial
* Untreated or insufficiently treated thyriodale disorders (if the patient is stable in the opinion of the physician, he may participate in the study)
* Cardiac edema
* Participation in weight reduction programs in the past 30 days
* Patients with swallowing problems, intestinal polyps or severe digestive disorders
* Patients with a history of constipation
* Patients who take drugs containing fat-soluble active substances and in which the time-consuming conditions of these drugs (see instructions for taking in Appendix O) are incompatible with the intake instructions of this study.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 165 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-04-16 (Actual)

PRIMARY OUTCOMES:
Changes in Bodyweight | Every two weeks (Start, 2 weeks, 4 weeks, 6 weeks, 8 Weeks)
  Changes in bodyweight during the study (weight reduction in kg). Comparison of the values obtained on day1 with results from day 65.

SECONDARY OUTCOMES:
Changes in BMI | Every two weeks (Start, 2 weeks, 4 weeks, 6 weeks, 8 Weeks)
  Changes in body-mass-index during the study. Comparison of the values obtained on day1 with results from day 65.
Safety: occurence of adverse events | Every week (from week 1 to week 10)
  Explore the occurence of adverse Events in the three different arms.
Changes in blood pressure | Every two weeks (Start, 2 weeks, 4 weeks, 6 weeks, 8 Weeks)
  Changes in blood pressure values during the study. Comparison of the values obtained on day1 with results from day 65.

CONTACTS AND LOCATIONS:
Locations (1):
- MIT Gesundheit GmbH, Kleve, North Rhine-Westphalia, Germany